CLINICAL TRIAL: NCT06411990
Title: Laser In Situ Fenestration for Endovascular Aortic Repair (LIFE) Study
Brief Title: Laser In Situ Fenestration Study
Acronym: LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Bath (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor-Investigator, Jonathan Bath, Associate Professor of Surgery, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2102631; 2023-001 (Other: University of Missouri)
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Aortic Aneurysm; Endovascular Aneurysm Repair
Keywords: Fenestrated Endovascular Aneurysm Repair
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: Prospective, single arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Endovascular Aneurysm Repair (Experimental): Fenestrated Endovascular Aneurysm Repair using the LIFE Device System
  Interventions: Device: Fenestrated Endovascular Aneurysm Repair using the LIFE Device System

INTERVENTIONS:
Device: Fenestrated Endovascular Aneurysm Repair using the LIFE Device System — Fenestrated Endovascular Aneurysm Repair
  Other Names: Medtronic Valiant Thoracic Stent Graft with the Captive Delivery System; Medtronic Endurant II Stent Graft System; Medtronic Endurant IIs Stent Graft System and/or; Medtronic Endurant Aorto-uni-iliac (AUI) Stent Graft System; GORE VIABAHN VBX Balloon Expandable Endoprostheses; Spectranetics CVX-300 Excimer Laser System with the Spectranetics Turbo-Elite Laser Atherectomy Catheter

SUMMARY:
The goal of this clinical trial is to learn about a new device, named the LIFE device, to treat people with aneurysms (swellings) in the aorta (large, main blood vessel that delivers blood from the heart to the body). The main questions this trial aims to answer are:

* If the LIFE device works to treat aortic aneurysms
* What medical problems participants have when the LIFE device is used Participants will undergo treatment with the LIFE device and thereafter at 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years have their pulses checked, bloodwork to check kidney function (BUN and serum creatinine), and a CT scan of the aneurysm area.

DETAILED DESCRIPTION:
In this clinical trial the LIFE device is used to treat people with aneurysms in the aorta near the kidney arteries (called juxtarenal or pararenal aortic aneurysms). Tubes, called stent grafts, are typically inserted through blood vessels in the groin and placed inside the aorta in the abdomen and chest area (endovascularly placed) to cover the tear or leak in the aorta. The LIFE device covers the tear or leak and has side branches to let blood flow into the kidney, spleen, intestine, or liver arteries. Participants in this study are not candidates for endovascular devices approved for endovascular aorta repair to the juxtarenal or pararenal aorta, not candidates for open repair, not willing to travel to sites that have access to manufacturer-made endovascular devices, and patients for whom there are no favorable alternatives, for example, urgent, symptomatic, and emergency cases.

ELIGIBILITY:
Inclusion Criteria:

1. Aortic aneurysm >5.5 cm in a man or > 5.0 cm in a woman or rapid expansion deemed at significant risk for rupture in the juxtarenal or pararenal aorta.
2. Endovascular aortic repair requiring coverage of renovisceral branches.
3. Not candidate or at high risk for open repair. For example, but not exclusively, due to renal dysfunction, previous abdominal surgery, obese body habitus, previous coronary bypass grafts or high cardiac risk, chronic obstructive pulmonary disease (COPD) or on oxygen at rest, poorly controlled diabetes, current smoking, or antiplatelet or anticoagulation use.
4. Proximal aortic landing zone in Zone 5 of the aorta or previous graft of at least 10 mm in length and diameter of between 20 and 40 mm.
5. Distance ≥ 5 mm between top of graft fabric and renovisceral branch orifice.
6. At least a 5 mm iliofemoral artery to accept the endovascular stent graft device and an axillary brachial artery of sufficient diameter to accept the laser catheter.
7. Renovisceral diameter between 4 and 13 mm at the origin.
8. At the time of case planning, the patient's anatomy appears amenable to complete exclusion of the aneurysm with laser fenestration techniques.
9. Not willing or able to travel to sites that have access to manufacturer-made investigational endovascular devices.
10. Not a candidate for currently approved endovascular options.
11. 18 years or older.
12. Patient or legally authorized representative agrees to participate in the study and provides written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.
13. Patient is able and willing to meet all study requirements, including participating in follow up evaluations and attending required assessment visits.

Exclusion Criteria:

1. Known sensitivities or allergies to the materials of construction of the devices, including Nitinol, polyester, Platinum-Iridium, stainless steel, fluoropolymer, and heparin.
2. Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed.
3. Uncorrectable coagulopathy.
4. Body habitus that would inhibit radiographic visualization of the aorta or exceeds the safe capacity of equipment.
5. Concurrent participation in another research protocol for investigation of an experimental therapy.
6. Subject has been judged to be unsuitable for participation in the study by the Investigator for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with freedom from death and major adverse events (MAE) | 30 days
  Number of subjects with freedom from all cause mortality and freedom from major adverse events. Major adverse events include myocardial infarction, chronic renal insufficiency / chronic renal failure requiring, dialysis, bowel ischemia, stroke, paraplegia or paraparesis, and prolonged ventilatory support.
Number of participants with device procedure technical success and freedom from endoleak, migration, aortic enlargement, aortic rupture, and aortic or branch-related reinterventions in | 12 months
  Device technical success (at the end of index procedure) and freedom from Type I and III endoleak, device migration ≥ 10 mm, aortic enlargement ≥ 5 mm, aortic rupture, and aortic or branch-related reinterventions, including conversion to open repair (within 12 months of the index procedure)

SECONDARY OUTCOMES:
Number of participants with delivery and deployment of the LIFE Device System | Procedure
  Ability to deliver and deploy the LIFE Device System
Number of participants with delivery and deployment of the thoracic/abdominal stent graft | Procedure
  Ability to deliver and deploy the thoracic/abdominal stent graft
Number of participants with coverage of intended aneurysm | Procedure
  Ability to cover the intended aneurysm
Number of participants with contrast flow into target renovisceral vessels | Procedure
  Contrast flow into the target renovisceral vessels
Estimated blood loss | Procedure
  Estimated blood loss
Ventilator days | From Procedure until the date of Hospital Discharge, typically 1-2 days
  Ventilator days
Days to oral intake | From Procedure until the date of Hospital Discharge, typically 1-2 days
  Days to oral intake
Intensive Care Unit (ICU) days | From Procedure until the date of Hospital Discharge, typically 1-2 days
  ICU days recorded
Days to hospital discharge | From Procedure until the date of Hospital Discharge, typically 1-2 days
  Days to hospital discharge
Procedure time | Procedure
  Procedure time (minutes)
Fluoroscopy time | Procedure
  Fluoroscopy time (minutes)
Endoleak rate | 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
  Endoleak rate at 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
Number of participants with device integrity failure | 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
  Device integrity failure (e.g., fracture) at 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
Number of participants with branch vessel device events | 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
  Branch vessel device events (i.e., kink, stenosis, or occlusion at 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
Number of participants with aortic growth | 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
  Aortic growth - defined as an increase ≥ 5 mm in maximal aortic diameter in any segment at 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
Number of participants with unplanned secondary procedures | 5 Years
  Unplanned secondary procedures throughout follow-up (e.g., unanticipated aortic or branch-related reoperation)
Number of participants with device migration | 6 Months, and 1, 2, 3, 4, and 5 Years
  Device migration (radiographic), antegrade or retrograde movement of more than 10 mm relative to anatomic landmarks identified on the first (30 Day) post-operative CT scan, at 6 Months, and 1, 2, 3, 4, and 5 Years
All adverse events | 5 Years
  All adverse events throughout 5 year follow-up, including if MAE, serious adverse event (SAE) or unanticipated adverse device effect (UADE), and the relationship of the AE to the LIFE Procedure and LIFE Device System
Freedom from aneurysm-related mortality | 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
  Freedom from aneurysm-related mortality at 30 Days, 6 Months, and 1, 2, 3, 4, and 5 Years
Freedom from all-cause mortality | 6 Months and 1, 2, 3, 4, and 5 Years
  Freedom from all-cause mortality at 6 Months and 1, 2, 3, 4, and 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bath, MD, Principal Investigator — University of Missouri School - Columbia
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No